CLINICAL TRIAL: NCT03687996
Title: Pratical Assessment of Descemet'Sstripping Automated Endothelial Keratoplasty (DSAEK) in the Management of Endothelial Decompensation Following Penetrating Keratoplasty
Brief Title: Pratical Assessment of DSAEK in the Management of Endothelial Decompensation Following Penetrating Keratoplasty
Acronym: MADE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-15Obs-CHRMT
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Descemet's Stripping Automated Endothelial Keratoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reporting our anatomical and functional results and the possible complications of the first six Descemet's stripping endothelial keratoplasty (DSAEK) performed in our department secondary to endothelial decompensation after penetrating keratoplasty.

DETAILED DESCRIPTION:
A retrospective and observational monocentric study fo six patients with DSAEK after prior penetrating keratoplasty (PK). The data collected are: demographic characteristics, ophthalmological comorbidities, initial indication of PK, delay between PK and DSAEK. Preoperative Visual Acuity and at 1, 3 and 6 months postoperative were collected in logmar for analysis. The central cornea and graft thickness measured in OCT as well as the postoperative complications were also collected.

ELIGIBILITY:
Inclusion Criteria:

* with endothelial decompensation after penetrating keratoplasty
* surgery realised by the same surgeon

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who profited of the first Descemet's stripping endothelial keratoplasty to endothelial decompensation after penetrating keratoplasty
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
visual acuity | change from visual acuity at 6 month
  pre and postoperative visual acuity in logmar

SECONDARY OUTCOMES:
cornea thickness at 6 months | change from cornea thickness at 6 months
  the central cornea and graft thickness measured in OCT
cornea thickness at 10 years | change from cornea thickness at 10 years
  the central cornea and graft thickness measured in OCT
postoperative complications | month 6
  all the postoperative complications were collected
visual acuity at 10 years | change from visual acuity at 10 years
  pre and postoperative visual acuity in logmar